CLINICAL TRIAL: NCT00885885
Title: An Open Label Randomized, Multi-Centre Exploratory Phase II Study to Evaluate the Efficacy and Safety of the Combination of Panitumumab With FOLFOX 4 Chemotherapy or Panitumumab With FOLFIRI Chemotherapy in Subjects With Wild- Type KRAS Colorectal Cancer and Liver-only Metastases.
Brief Title: Safety and Efficacy Study of FOLFOX4+Panitumumab vs.FOLFIRI+Panitumumab in Subjects WT KRAS Colorectal Cancer and Liver-only Metastases
Acronym: PLANET
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Spanish Cooperative Group for the Treatment of Digestive Tumours (TTD) (Other)
Collaborators: Amgen (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TTD-08-04; EudraCT: 2008-006766-28
Record Dates: First submitted 2009-04-21; First posted 2009-04-22 (Estimated); Last update posted 2017-08-01 (Actual); Status verified 2017-07

CONDITIONS: Colorectal Cancer
Keywords: Colorectal Cancer; Panitumumab; FOLFOX-4; FOLFIRI
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): Panitumumab+FOLFOX 4
  Interventions: Drug: Panitumumab+FOLFOX-4
- 2 (Experimental): Panitumumab+FOLFIRI
  Interventions: Drug: Panitumumab+FOLFIRI

INTERVENTIONS:
Drug: Panitumumab+FOLFOX-4 — Panitumumab will be administered as a 60-minute ± 15 minutes IV infusion, just prior to administration of chemotherapy at a dose of 6 mg/kg on day 1 of each cycle. If the first infusion of panitumumab is well tolerated (without any serious infusion related reactions) all subsequent infusions may be administered over 30 minutes ± 10 minutes.
  A cycle of panitumumab is defined as 14 days.
  FOLFOX 4 chemotherapy will be administered on day 1 of each 14-day treatment cycle:
  * Oxaliplatin 85mg/m2 as a 120 minute infusion on day 1 of each cycle
  * Folinic acid 200mg/m2 as a 120 minute infusion on days 1 and 2
  * A bolus (2 to 4 minutes) of 5-FU at 400mg/m2 on days 1 and 2
  * 5-FU at 600mg/m2 as a continuous infusion of 22 hour infusion on days 1 and 2
  Arms: 1
Drug: Panitumumab+FOLFIRI — Panitumumab will be administered as a 60-minute ± 15 minutes IV infusion, just prior to administration of chemotherapy at a dose of 6 mg/kg on day 1 of each cycle. If the first infusion of panitumumab is well tolerated (without any serious infusion related reactions) all subsequent infusions may be administered over 30 minutes ± 10 minutes.
  A cycle of panitumumab is defined as 14 days.
  FOLFIRI chemotherapy will be administered on day 1 of each 14-day treatment cycle:
  * Irinotecan 180 mg/m2 will be administered over 90 minutes ± 15 minutes on day 1 of each cycle
  * Folinic acid 400 mg/m2 will be administered over 2 hours ± 15 minutes during the irinotecan infusion but without mixing
  * A bolus (2 to 4 minutes) of 5-FU at 400mg/m2 on day 1
  * 5-FU at 2400 mg/m2 continuous intravenous infusion over 46-hour ± 2-hour on day 1 of each cycle.
  Arms: 2

SUMMARY:
The purpose of the study is to evaluate the efficacy and safety of the combination of Panitumumab with FOLFOX 4 Chemotherapy or Panitumumab with FOLFIRI Chemotherapy in Subjects with Wild- Type KRAS Colorectal Cancer and liver-only Metastases.

ELIGIBILITY:
Inclusion Criteria:

* Man or woman > 18 years < 75 of age
* Competent to comprehend, sign, and date an IEC-approved informed consent form
* Histologically confirmed adenocarcinoma of the colon or rectum
* Wild Type KRAS status
* Metastatic colorectal carcinoma exclusively affecting only the liver, compliant with one of the following criteria

  1. Number of liver metastasis ≥ 4.
  2. Size of one liver metastasis > 10 cm in diameter.
  3. Liver metastases technically not resectable.
* At least 1 uni-dimensionally measurable lesion
* Patients with the following characteristics will be included:

  1. Recurrence after adjuvant treatment with 5-fluorouracil/folinic acid or capecitabine +/- radiotherapy with a disease-free interval > than 6 months after its completion; or after oxaliplatin containing adjuvant treatment with a disease-free interval > than 12 months
  2. Recurrence after surgical treatment and/or radiotherapy with no adjuvant systemic treatment.
  3. De novo diagnosis of the disease.
* Patients with simultaneous liver metastases are eligible, if the primary tumor has been resected at least 1 month prior chemotherapy.
* Prior radiotherapy is acceptable.
* Patients deemed to have no major contra-indication to liver surgery from a general health perspective.
* Karnofsky performance status ≥ 70%
* Adequate bone marrow function: neutrophils ≥ 1.5 x109/ L; platelets ≥ 100 x109/ L;hemoglobin ≥ 9g/ dL
* Hepatic and metabolic function as follows:

Total bilirubin count ≤ 1.5 x ULN and not increasing more than 25% within the last 4 weeks; ALAT and ASAT < 5 x ULN;

* Renal function, calculated creatinine clearance or 24 hour creatinine clearance ≥ 50 mL/ min.
* Magnesium > LLN

Exclusion Criteria:

* Prior anti-EGFr antibody therapy (eg, cetuximab) or treatment small molecule EGFr tyrosine kinase inhibitors (eg, erlotinib).Subjects who have experienced an infusion reaction to their first dose of anti-EGFR therapy (cetuximab) may participate in this clinical trial.
* Surgery (not including diagnostic biopsy) and/or radiotherapy in the 4 weeks prior to inclusion in the study.
* Metastasis on any site other than the liver, including extrahepatic lymph nodes.
* Prior malignant tumor in the last 5 years, except a history of basal cell carcinoma of the skin or pre-invasive carcinoma of the skin.
* Systemic chemotherapy, hormonal therapy, immunotherapy or experimental or approved proteins/antibodies (eg, bevacizumab) ≤ 30 days before inclusion
* Unresolved toxicities from prior systemic therapy that, in the opinion of the investigator, does not qualify the patient for inclusion
* Significant cardiovascular disease including unstable angina or myocardial infarction within 6 months before initiating study treatment or a history of ventricular arrhythmia
* History of interstitial pneumonitis or pulmonary fibrosis or evidence of interstitial pneumonitis or pulmonary fibrosis on baseline chest CT scan
* Treatment for systemic infection within 14 days before initiating study treatment
* Active inflammatory bowel disease or other bowel disease causing chronic diarrhoea (defined as > 4 loose stools per day)
* History of Gilbert's syndrome or dihydropyrimidine deficiency
* History of any medical condition that may increase the risks associated with study participation or may interfere with the interpretation of the study results
* Known positive test for human immunodeficiency virus infection, hepatitis C virus, chronic active hepatitis B infection
* subject allergic to the ingredients of the study medication or to Staphylococcus protein A
* Any co-morbid disease that would increase risk of toxicity
* Any kind of disorder that compromises the ability of the subject to give written informed consent and/or comply with the study procedures
* Any investigational agent within 30 days before enrolment
* Must not have had a major surgical procedure within 28 days of randomization
* Subject who is pregnant or breast feeding
* Woman or man of childbearing potential not consenting to use adequate contraceptive precautions i.e. double barrier contraceptive methods (eg diaphragm plus condom), or abstinence during the course of the study and for 6 months after the last study drug administration for women, and 1 month for men
* Subject unwilling or unable to comply with study requirements

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2009-05; Primary Completion 2015-03 (Actual); Study Completion 2015-03 (Actual)

PRIMARY OUTCOMES:
Objective response rate | 2009-2013

SECONDARY OUTCOMES:
% of patients whose disease becomes resectable | 2009-2013
Time to resection | 2009-2013
Duration of response | 2009-2013
Progression-free survival | 2009-2013
Time to treatment failure | 2009-2013
Time to disease relapse following surgery. | 2009-2013
Adverse Events | 2009-2013
Evaluation of molecular predictive markers for response. | 2009-2013

CONTACTS AND LOCATIONS:
Overall Officials: Albert Abad, MD, phD, Study Chair — ICO-H. Germans Trial i Pujol. Badalona. Spain; Alfredo Carrato, MD, phD, Study Chair — Hospial Ramón y Cajal. Madrid. Spain
Locations (1):
- Spanish Cooperative Group for Gastrointestinal Tumour Therapy, Madrid, Spain

REFERENCES:
- [Derived] Benavides M, Diaz-Rubio E, Carrato A, Abad A, Guillen C, Garcia-Alfonso P, Gil S, Cano MT, Safont MJ, Gravalos C, Manzano JL, Sanchez A, Alcaide J, Lopez R, Massuti B, Sastre J, Martinez E, Escudero P, Mendez M, Aranda E. Tumour location and efficacy of first-line EGFR inhibitors in KRAS/RAS wild-type metastatic colorectal cancer: retrospective analyses of two phase II randomised Spanish TTD trials. ESMO Open. 2019 Dec 1;4(6):e000599. doi: 10.1136/esmoopen-2019-000599. eCollection 2019. PMID 31803504
- [Derived] Carrato A, Abad A, Massuti B, Gravalos C, Escudero P, Longo-Munoz F, Manzano JL, Gomez A, Safont MJ, Gallego J, Garcia-Paredes B, Pericay C, Duenas R, Rivera F, Losa F, Valladares-Ayerbes M, Gonzalez E, Aranda E; Spanish Cooperative Group for the Treatment of Digestive Tumours (TTD). First-line panitumumab plus FOLFOX4 or FOLFIRI in colorectal cancer with multiple or unresectable liver metastases: A randomised, phase II trial (PLANET-TTD). Eur J Cancer. 2017 Aug;81:191-202. doi: 10.1016/j.ejca.2017.04.024. Epub 2017 Jun 19. PMID 28633089
- See also: Related Info — http://www.ttdgroup.org